CLINICAL TRIAL: NCT02542605
Title: Phase I, Randomized, Parallel-group, Double-Blind, Placebo-Controlled, Single Dose Study to Evaluate the Blockade of CGRP Receptor by AMG 334 in Preventing PACAP-38 Induced Migraine-like Attacks in Migraine Patients
Brief Title: To Evaluate the Blockade of CGRP in Preventing PACAP-38 Induced Migraine-like Attacks With AMG 334 in Migraine Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20140207
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Migraine
Keywords: Migraine; Headache; Migraine Headache; Headache, Migraine; Amgen
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab; Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PACAP-38 Challenge Agent (Other): In Part A, 4 cohorts of 2 to 5 participants sequentially received an intravenous infusion of 10 picomol/kilogram/minute (pmol/kg/minute) PACAP-38 for 2.5, 5, 7.5 and 10 minutes each in order to determine the dose for Part B.
  Interventions: Drug: PACAP-38 Challenge Agent
- Placebo (Placebo Comparator): Participants were randomized to receive matching erenumab placebo by intravenous administration over 30 minutes on day 1. On day 8 participants were administered the dose of PACAP-38 determined from Part A of the study (100 pmol/kg) and were followed up for 11 weeks.
  Interventions: Drug: Placebo; Drug: PACAP-38 Challenge Agent
- Erenumab (Experimental): Participants were randomized to receive 140 milligrams (mg) erenumab by intravenous administration over 30 minutes on day 1 in Part B. On day 8 participants were administered the dose of PACAP-38 determined from Part A of the study (100 pmol/kg) and were followed up for 11 weeks.
  Interventions: Drug: Erenumab; Drug: PACAP-38 Challenge Agent

INTERVENTIONS:
Drug: Erenumab — Administered once on day 1 of Part B of the study by intravenous infusion.
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab
Drug: Placebo — Administered once on day 1 of Part B of the study by intravenous infusion.
  Arms: Placebo
Drug: PACAP-38 Challenge Agent — Administered by intravenous infusion during Part A of the study for dose selection for Part B.
  Administered by intravenous infusion on day 8 in Part B as a challenge agent to induce a migraine-like attack.
  Other Names: Pituitary adenylate cyclase-activating polypeptide-38 (PACAP-38)

SUMMARY:
Phase I, Randomized, Parallel-group, Double-Blind, Placebo-Controlled, Single Dose Study to Evaluate the Blockade of CGRP Receptor by AMG 334 in Preventing PACAP-38 Induced Migraine-like Attacks in Migraine Patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 to ≤ 45 years of age upon entry into screening
* History of migraine headaches without aura for ≥ 6 months prior to screening according to the International Headache Society (IHS) International Classification of Headache Disorders (ICHD-II) (Headache Classification Committee of the International Headache Society, 2004) based on medical records and/or patient self-report
* Migraine frequency: ≥ 1 and ≤ 5 migraine days per month in each of the 3 months prior to screening

Exclusion Criteria:

* History of migraine with aura, cluster headache or hemiplegic migraine headache according to the IHS Classification ICHD-II (Headache Classification Committee of the International Headache Society, 2004) based on medical records and/or patient self-report
* ≥ 6 migraine days per month in the last 3 months prior to study enrollment and during screening period
* Other headache disorders (except for episodic tension-type headache <5 days/month)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- Research Site, Anaheim, California, United States
- Research Site, Leuven, Belgium
- Research Site, Leiden, Netherlands

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 2 centers in Belgium and the Netherlands from November 2015 until November 2017 when the study was terminated early due to slow recruitment rate. Additionally, 2 participants were enrolled at a center in the United States for Part A prior to this study site being closed.
Pre-assignment Details: 12 participants received treatment in Part A to determine the lowest pituitary adenylate cyclase-activating polypeptide-38 (PACAP-38) dose that triggered a migraine-like attack (MLA). PACAP-38 responders from Part A and PACAP-38 naïve participants were randomized in Part B (17 in total). 35 participants were enrolled in the study (Parts A and B).
Groups:
- PACAP-38 Challenge Agent: In Part A, cohorts 1 to 4 (of 2 to 5 participants each) sequentially received an intravenous infusion of 10 picomol/kilogram/minute (pmol/kg/minute) PACAP-38 over 2.5, 5, 7.5 and 10 minutes, respectively. Dose selection in Part A enabled the dose for Part B to be determined.
  PACAP-38 naïve participants entered the study at Part B. On day 1 of the Part B challenge phase participants received the dose of PACAP-38 determined from Part A of the study: 100 pmol/kg (administered as 10 pmol/kg/minute PACAP-38 over 10 minutes). Responders who experienced a MLA within 24 hours were screened for the randomization phase.
- Placebo: Participants were randomized to receive matching erenumab placebo by intravenous administration over 30 minutes on day 1 of Part B randomization phase. On day 8, participants were administered the dose of PACAP-38 determined from Part A of the study (100 pmol/kg) and were followed up for 11 weeks.
- Erenumab: Participants were randomized to receive 140 milligrams (mg) erenumab by intravenous administration over 30 minutes on day 1 of Part B randomization phase. On day 8, participants were administered the dose of PACAP-38 determined from Part A of the study (100 pmol/kg) and were followed up for 11 weeks.
Period: Part A: PACAP-38 Dose Selection Phase
Arm/Group | PACAP-38 Challenge Agent | Placebo | Erenumab
Started | 12 | 0 | 0
Received PACAP-38 | 12 | 0 | 0
Proceeded to Part B Randomization Phase | 2 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part B: Challenge Phase
Arm/Group | PACAP-38 Challenge Agent | Placebo | Erenumab
Started (Participants starting Part B are all PACAP-38 naïve and did not participate in Part A.) | 23 | 0 | 0
Received PACAP-38 | 23 | 0 | 0
Proceeded to Randomization Phase | 15 | 0 | 0
Completed | 22 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 0 | 0
Period: Part B: Randomization Phase
Arm/Group | PACAP-38 Challenge Agent | Placebo | Erenumab
Started | 0 | 9 | 8
Not PACAP-38 naïve Participants (Participants received PACAP-38 during Part A dose selection.) | 0 | 2 | 0
PACAP-38 naïve Participants (Participants joined the study at Part B and did not receive PACAP-38 in Part A.) | 0 | 7 | 8
Received Placebo/Erenumab | 0 | 9 | 7
Completed | 0 | 9 | 7
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall baseline population consists of all participants who received at least 1 dose of PACAP-38 in either Part A or Part B of the study.
Groups:
- PACAP-38 Challenge Agent: In Part A, cohorts 1 to 4 (of 2 to 5 participants each) sequentially received an intravenous infusion of 10 pmol/kg/minute PACAP-38 over 2.5, 5, 7.5 and 10 minutes, respectively. Dose selection in Part A enabled the dose for Part B to be determined.
  PACAP-38 naïve participants entered the study at Part B. On day 1 of the Part B challenge phase participants received the dose of PACAP-38 determined from Part A of the study: 100 pmol/kg (administered as 10 pmol/kg/minute PACAP-38 over 10 minutes). Responders who experienced a MLA within 24 hours were screened for the randomization phase.
Arm/Group | PACAP-38 Challenge Agent
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (6.2)
Age, Customized [Number; unit: Participants]
  18 - 64 years | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3
  Black (or African American) | 2
  Multiple (Asian-White) | 1
  White | 28
  Other | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
Height [Mean (Standard Deviation); unit: centimeters] | 168.13 (7.72)
Weight [Mean (Standard Deviation); unit: kg] | 69.433 (14.656)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.4738 (4.2926)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a MLA Within 24 Hours of Challenge Agent Infusion
Description: On day 1 of the double-blind randomization phase participants received 140 mg intravenous erenumab over 30 minutes or matching placebo. On day 8, participants received 10 mol/kg/minute PACAP-38 over 10 minutes and were observed for 24 hours after PACAP-38 infusion.
  A MLA was defined as fulfilling 1 of the 2 criteria:
  1. Headache with at least 2 of the following characteristics: unilateral location, pulsating quality, moderate or severe pain intensity, aggravated by/causing avoidance of routine physical activity. Additionally, during the headache at least 1 of the following: nausea and/or vomiting, photophobia or phonophobia.
  2. Headache described as mimicking usual migraine attack treated with triptan.
Time Frame: Part B randomization phase day 8 plus 24 hours.
Population: The Safety Analysis Set consisted of all randomized participants who received at least 1 dose of investigational product (placebo or erenumab) in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Erenumab: Participants were randomized to receive 140 mg erenumab by intravenous administration over 30 minutes on day 1 of Part B randomization phase. On day 8, participants were administered the dose of PACAP-38 determined from Part A of the study (100 pmol/kg) and were followed up for 11 weeks.
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants
  Participants with MLA | 1 | 1
  Participants without MLA | 8 | 6

2. Secondary Outcome: Number of Participants With a Headache Within 24 Hours of Challenge Agent Infusion
Description: On day 1 of the double-blind randomization phase participants received 140 mg intravenous erenumab over 30 minutes or matching placebo. On day 8, participants received 10 mol/kg/minute PACAP-38 over 10 minutes and were observed for 24 hours after PACAP-38 infusion.
Time Frame: Part B randomization phase day 8 plus 24 hours.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants
  Participants with headaches | 3 | 3
  Participants without headaches | 6 | 4

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were summarised for days 1 to 7 after the participants received placebo or erenumab infusion on day 1 of the Part B randomization phase. TEAEs were also summarized from day 8 to end of study (EOS) after participants had received both investigational product (placebo or erenumab) and the second dose of PACAP-38 on day 8.
Time Frame: Part B randomization phase day 1 until EOS (up to 12 weeks).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants
  Participants with TEAEs from day 1 to 7 | 6 | 0
  Participants with TEAEs from day 8 to EOS | 9 | 7
  Serious AEs | 0 | 0
  AEs with fatal outcome | 0 | 0

4. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at Day 1, Day 8 and EOS
Description: Systolic and diastolic BP was assessed during Part B of the study, and the mean change from baseline is presented for the last measurements taken following administration of placebo or erenumab on day 1 (1 hour post-dose), and following administration of PACAP-38 on day 8 (8 hours post-dose). The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization phase baseline and day 1, day 8 and EOS (week 12).
Population: The Safety Analysis Set consisted of all randomized participants who received at least 1 dose of investigational product (placebo or erenumab) in Part B. Only participants with data available for analysis at each time point are presented.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
millimeters of mercury
  1 hour post-dose day 1: systolic BP | -0.7 (7.9) | 2.4 (5.2)
  1 hour post-dose day 1: diastolic BP | 1.2 (5.7) | 0.7 (6.4)
  8 hours post-dose day 8: systolic BP: number analyzed (Participants) | 8 | 7
  8 hours post-dose day 8: systolic BP | -3.1 (5.7) | -3.7 (6.2)
  8 hours post-dose day 8: diastolic BP: number analyzed (Participants) | 8 | 7
  8 hours post-dose day 8: diastolic BP | -3.6 (2.9) | -9.6 (6.8)
  EOS: systolic BP | -2.6 (9.2) | 2.6 (3.8)
  EOS: diastolic BP | -0.1 (6.4) | 1.7 (5.9)

5. Secondary Outcome: Mean Change From Baseline in Heart Rate at Day 1, Day 8 and EOS
Description: Heart rate was assessed during Part B of the study, and the mean change from baseline is presented for the last measurements taken following administration of placebo or erenumab on day 1 (1 hour post-dose), and following administration of PACAP-38 on day 8 (8 hours post-dose). The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization phase baseline and day 1, day 8 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
beats/minute
  1 hour post-dose day 1 | -5.0 (8.2) | 1.7 (5.7)
  8 hours post-dose day 8: number analyzed (Participants) | 8 | 7
  8 hours post-dose day 8 | 2.6 (11.5) | 8.7 (4.6)
  EOS | -0.9 (8.6) | 2.4 (5.5)

6. Secondary Outcome: Mean Change From Baseline in Respiratory Rate at Day 1, Day 8 and EOS
Description: Respiratory rate was assessed during Part B of the study, and the mean change from baseline is presented for the last measurements taken following administration of placebo or erenumab on day 1 (1 hour post-dose), and following administration of PACAP-38 on day 8 (8 hours post-dose). The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization phase baseline and day 1, day 8 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
breaths/minute
  1 hour post-dose day 1 | 0.8 (2.2) | -1.4 (2.6)
  8 hours post-dose day 8: number analyzed (Participants) | 8 | 7
  8 hours post-dose day 8 | 1.0 (2.1) | -1.0 (3.5)
  EOS | 1.7 (4.0) | 1.1 (3.7)

7. Secondary Outcome: Mean Change From Baseline in Temperature at Day 1, Day 8 and EOS
Description: Temperature was assessed during Part B of the study, and the mean change from baseline is presented for the last measurements taken following administration of placebo or erenumab on day 1 (1 hour post-dose), and following administration of PACAP-38 on day 8 (8 hours post-dose). The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization phase baseline and day 1, day 8 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
degrees Celsius
  1 hour post-dose day 1 | 0.18 (0.39) | 0.34 (0.36)
  8 hours post-dose day 8: number analyzed (Participants) | 8 | 7
  8 hours post-dose day 8 | 0.60 (0.48) | 0.63 (0.56)
  EOS | -0.34 (0.47) | 0.16 (0.41)

8. Secondary Outcome: Mean Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) at Day 8, Day 9 and EOS
Description: ALP, ALT and AST were assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization phase baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Units/Liter
  Day 8 (Pre-PACAP-38 dose): ALP: number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose): ALP | -2.0 (5.6) | 0.0 (4.8)
  Day 9 (Post-PACAP-38 dose): ALP: number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose): ALP | -1.6 (4.1) | -0.3 (2.3)
  EOS: ALP | 1.0 (12.3) | 6.1 (9.6)
  Day 8 (Pre-PACAP-38 dose): ALT: number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose): ALT | -1.4 (3.5) | -3.0 (4.2)
  Day 9 (Post-PACAP-38 dose): ALT: number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose): ALT | -2.1 (3.5) | -4.5 (4.2)
  EOS: ALT | -2.0 (4.7) | 3.1 (9.4)
  Day 8 (Pre-PACAP-38 dose): AST: number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose): AST | 0.3 (3.0) | 2.4 (4.0)
  Day 9 (Post-PACAP-38 dose): AST: number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose): AST | -0.8 (2.7) | -4.2 (2.3)
  EOS: AST | 0.3 (5.1) | -0.4 (3.6)

9. Secondary Outcome: Mean Change From Baseline in Total Bilirubin at Day 8, Day 9 and EOS
Description: Total bilirubin was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
micromol/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 7 | 7
  Day 8 (Pre-PACAP-38 dose) | -0.4211 (3.6356) | -1.4849 (0.8532)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 7 | 6
  Day 9 (Post-PACAP-38 dose) | 3.3229 (1.3971) | -2.2980 (1.0300)
  EOS: number analyzed (Participants) | 8 | 7
  EOS | 0.0804 (3.0270) | 1.3191 (3.5099)

10. Secondary Outcome: Mean Change From Baseline in Blood Urea at Day 8, Day 9 and EOS
Description: Blood urea was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimol/L (mmol/L)
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
millimol/L (mmol/L)
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | 0.0629 (0.9274) | -0.0524 (0.5270)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | 0.1501 (0.7552) | -0.5278 (1.2592)
  EOS | -0.1961 (0.7673) | 0.0570 (1.1286)

11. Secondary Outcome: Mean Change From Baseline in Creatine Kinase at Day 8, Day 9 and EOS
Description: Creatine Kinase was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
U/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | 5.8 (21.0) | -22.4 (51.5)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | -16.8 (9.1) | -59.3 (65.7)
  EOS | 8.1 (25.3) | -24.9 (79.9)

12. Secondary Outcome: Mean Change From Baseline in Creatinine at Day 8, Day 9 and EOS
Description: Creatinine was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
micromol/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | -1.9890 (6.0835) | -2.2526 (3.1121)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | 0.1450 (7.3859) | -1.4733 (3.4367)
  EOS | 3.5151 (7.8109) | -0.3457 (2.6598)

13. Secondary Outcome: Mean Change From Baseline in Direct Bilirubin at Day 8, Day 9 and EOS
Description: Direct bilirubin was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
micromol/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 3 | 1
  Day 8 (Pre-PACAP-38 dose) | -0.0570 (1.2948) | -1.0260 (NA) — Only 1 participant was analysed for this timepoint.
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 3 | 2
  Day 9 (Post-PACAP-38 dose) | 0.6270 (0.5497) | -1.1115 (0.1209)
  EOS: number analyzed (Participants) | 3 | 2
  EOS | 0.1710 (0.1710) | 1.1970 (0.0000)

14. Secondary Outcome: Mean Change From Baseline in Eosinophil Count at Day 8, Day 9 and EOS
Description: Eosinophil count was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
10^9/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | -0.013 (0.067) | -0.004 (0.046)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | -0.035 (0.076) | -0.002 (0.066)
  EOS | -0.041 (0.060) | 0.033 (0.061)

15. Secondary Outcome: Mean Change From Baseline in Blood Glucose at Day 8, Day 9 and EOS
Description: Blood glucose was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
mmol/L
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | -0.1360 (0.3103) | -0.2761 (0.5961)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | -0.2290 (0.2350) | 0.0427 (0.2432)
  EOS | -0.3183 (0.3395) | -0.1237 (0.3645)

16. Secondary Outcome: Mean Change From Baseline in Hemoglobin A1C (Fraction of 1) at Day 8, Day 9 and EOS
Description: Hemoglobin A1C was assessed during Part B of the study, and the mean change from baseline is presented for samples taken prior to administration of PACAP-38 on day 8 (pre-PACAP-38 dose), and following administration of PACAP-38 on day 9. The mean change from baseline is also presented for the EOS assessment.
Time Frame: Part B randomization baseline and day 8, day 9 and EOS (week 12).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: fraction of 1
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
fraction of 1
  Day 8 (Pre-PACAP-38 dose): number analyzed (Participants) | 8 | 7
  Day 8 (Pre-PACAP-38 dose) | 0.0003 (0.0007) | 0.0001 (0.0007)
  Day 9 (Post-PACAP-38 dose): number analyzed (Participants) | 8 | 6
  Day 9 (Post-PACAP-38 dose) | 0.0000 (0.0005) | 0.0002 (0.0010)
  EOS: number analyzed (Participants) | 9 | 6
  EOS | 0.0003 (0.0012) | 0.0002 (0.0012)

17. Secondary Outcome: Pharmacokinetics (PK): Mean Erenumab Serum Concentration at 1 Hour (C1h)
Description: The mean serum erenumab concentration at 1 hour post-dose on day 1 of Part B randomization phase is presented.
Time Frame: Part B randomization phase 1 hour post-dose day 1.
Population: The PK Analysis Set consisted of all randomized participants who received erenumab and have at least 1 PK concentration result.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Erenumab
Number analyzed (Participants) | 7
micrograms per milliliter (mcg/mL) | 51.2 (9.72)

18. Secondary Outcome: PK: Mean Area Under the Concentration-time Curve From Time 0 to 84 Days Post-dose (AUC84d)
Description: The mean AUC84d for erenumab for the Part B randomization phase is presented.
Time Frame: Part B randomization phase baseline and 84 days post-dose.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Erenumab
Number analyzed (Participants) | 7
day*mcg/mL | 877 (131)

19. Secondary Outcome: Number of Participants With Anti-Erenumab Antibodies
Description: Participants were tested for binding antibodies and neutralizing antibodies at baseline and following treatment with erenumab.
Time Frame: Part B randomization phase baseline and EOS.
Population: The Safety Analysis Set for erenumab consisted of all randomized participants who received at least 1 dose of erenumab in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab
Number analyzed (Participants) | 7
Participants
  Binding antibody positive at/before baseline | 0
  Neutralizing antibody positive at/before baseline | 0
  Binding antibody positive post-baseline | 0
  Neutralizing antibody positive post-baseline | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: At baseline, 12-lead ECGs were performed in a standardized method, in triplicate, and approximately 30 seconds apart, prior to blood draws or other invasive procedures. Single ECGs were performed from Day 1 to EOS. ECG results were reviewed by the investigator and classified as: normal, abnormal not clinically significant or abnormal, clinically significant. The number of participants with abnormal, clinically significant changes in ECG results at EOS are presented.
Time Frame: Part B randomization phase baseline and EOS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Parameters
Description: Physical examinations were performed by an investigator and any abnormal findings, judged to be clinically significant were recorded as an AE. The number of participants with clinically significant changes in physical parameters at EOS are presented.
Time Frame: Part B randomization phase baseline and EOS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Changes in Neurological Assessments
Description: Neurological examinations including assessment of cranial nerves, motor system, sensory system (including testing for pain sensation [pin prick], light touch sensation [brush], von Frey, and vibratory sense), reflexes, and cerebellar function were performed by the investigator and classified as normal or abnormal. Any abnormal findings, judged by the investigator to be clinically significant, were recorded as an AE. The number of participants with clinically significant changes in neurological assessments at EOS are presented.
Time Frame: Part B randomization phase baseline and EOS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of investigational product (placebo or erenumab) up to 85 days (up to 12 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of AEs that exceed the indicated frequency threshold.
Groups:
- Placebo Day 1-7: Participants were randomized to receive matching erenumab placebo intravenously over 30 minutes on study day 1 of Part B randomization phase.
- Erenumab Day 1-7: Participants were randomized to receive 140 mg erenumab intravenously over 30 minutes on study day 1 of Part B randomization phase.
- Placebo Day 8-EOS: On day 8 of Part B randomization phase, participants were administered 100 pmol/kg of PACAP-38, having received matching erenumab placebo on day 1. Participants were followed up for 11 weeks to EOS.
- Erenumab Day 8-EOS: On day 8 of Part B randomization phase, participants were administered 100 pmol/kg of PACAP-38, having received 140 mg erenumab intravenously on day 1. Participants were followed up for 11 weeks to EOS.
Arm/Group | Placebo Day 1-7 | Erenumab Day 1-7 | Placebo Day 8-EOS | Erenumab Day 8-EOS
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 6/9 | 0/7 | 9/9 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Day 1-7 (N=9) | Erenumab Day 1-7 (N=7) | Placebo Day 8-EOS (N=9) | Erenumab Day 8-EOS (N=7)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 5 | 5
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 2
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Catheter site pain (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 4 | 5
Feeling cold (General disorders) | 0 | 0 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 3 | 2
Hunger (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Thirst decreased (General disorders) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 4 | 1
Headache (Nervous system disorders) | 0 | 0 | 6 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 3 | 0 | 6 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 7 | 6

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow recruitment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02542605/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT02542605/SAP_001.pdf